CLINICAL TRIAL: NCT02427061
Title: Engendering Healthy Masculinities to Prevent Sexual Violence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Elizabeth Miller, Chief, Division of Adolescent and Young Adult Medicine, Children's Hospital, UPMC, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 14080673
Record Dates: First submitted 2015-04-17; First posted 2015-04-27 (Estimated); Last update posted 2018-07-23 (Actual); Status verified 2018-07

CONDITIONS: Violence; Sexual Assault

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Program (Manhood 2.0) (Experimental): Curricular Content: The 18 hour content will be spread over 3 to 6 sessions (3 weeks duration up to a 2 month period). Youth are guided to explore social constructions of masculinity, describe healthy relationships, discuss healthy sexual behaviors, identify coercive and disrespectful behaviors, and practice skills to intervene when witnessing peers' disrespectful and harmful behaviors, with repeated reflection on gender norms throughout these sessions.
  Module One focuses on themes of gender and masculinity. Module Two focuses on themes of violence and sexual consent. Module Three focuses on themes of sexual health and decision making.
  Interventions: Behavioral: Intervention Program (Manhood 2.0)
- Control Program (Job Skills Training) (Active Comparator): Youth in the control arm receive the same amount of time with an intervention -- 18 hours of curriculum divided into 3 to 6 sessions, over 3 weeks up to 2 months duration.
  The control intervention focuses on job skills development.
  Interventions: Behavioral: Control Program (Job Skills Training)

INTERVENTIONS:
Behavioral: Intervention Program (Manhood 2.0)
  Arms: Intervention Program (Manhood 2.0)
Behavioral: Control Program (Job Skills Training)
  Arms: Control Program (Job Skills Training)

SUMMARY:
Sexual violence (SV) and adolescent relationship abuse (ARA) are prevalent among adolescents and associated with poor health. Global health organizations highlight engaging men and boys in preventing violence against women as a potentially impactful public health strategy. This study aims to test, via a two arm cluster randomized controlled trial, a "gender transformative" SV/ARA perpetration prevention program among African American adolescent males ages 13-19 (target is high school age) implemented in a community-based setting. "Gender transformative" refers to a theory- and evidence-based approach to alter gender norms that foster SV/ARA while promoting bystander intervention (i.e., giving boys skills to interrupt abusive behaviors they witness among peers) to reduce SV/ARA perpetration. As the acceptance of SV and involvement in unhealthy sexual behaviors are associated with SV/ARA perpetration, this program integrates analysis of social norms that condone violence against women, sexual health promotion, and skills in bystander intervention -- an approach that has been implemented in multiple non-U.S. settings among young adult males with reductions in violence, development of more equitable gender attitudes, and less risky sexual behaviors. This will be the first test of such a gender transformative program among adolescent males in the U.S. Via a 2-arm cluster-randomized trial in youth-serving agencies (16 clusters, N=840 adolescent males ages 14-19), this study will assess the effectiveness of "Manhood 2.0" (proposed name for this gender transformative program) compared to a job skills curriculum. Three months after the end of the program (Time 2), compared to controls, youth will demonstrate increased positive bystander intervention behaviors (secondary outcome). Intermediate outcomes are: condom use self-efficacy; contraception use attitudes; recognition of abusive behaviors; gender-equitable attitudes; and intentions to intervene with peers. Nine months after intervention completion (Time 3), youth will report less perpetration of SV and ARA toward females (Primary Outcome) compared to controls. This study will provide urgently needed information about the effectiveness of a gender transformative program that combines healthy sexuality skills, gender norms change, and bystander skills to interrupt peers' disrespectful and harmful behaviors to reduce SV/ARA perpetration among adolescent males.

ELIGIBILITY:
Inclusion criteria:

* adolescent males ages 13-19
* recruited from youth-serving agencies in the Pittsburgh region
* able to provide their own assent
* English speaking

Exclusion criteria:

* adolescent males younger than 13 years old or older than 19 years old
* not able to provide their own assent
* non- English speaking

Ages: 13 Years to 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 868 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in self-reported perpetration of Sexual Violence and Adolescent Relationship Abuse at Time 3 | 9 months after intervention (Time 3)
  Assessment of Sexual Violence and Adolescent Relationship Abuse perpetration comparing baseline summary score with follow up summary score (whether they have perpetrated acts of Sexual Violence or Relationship Abuse towards anyone)

SECONDARY OUTCOMES:
Change in Positive Bystander Behavior from Baseline to Follow Up | 3 months after intervention (Time 2), 9 months after intervention (Time 3)
  Assessment of positive bystander behavior in participants over the past 3 months when witnessing disrespectful and harmful behavior among peers comparing baseline and follow up summary scores. Participants report if they have witnessed peers' abusive behaviors in the past 3 months and if witnessed, how they responded (whether they intervened to interrupt the behavior)

OTHER OUTCOMES:
Change in Intentions to Intervene from Baseline to Follow Up | 3 months after intervention (Time 2), 9 months after intervention (Time 3)
  Proclivity to intervene when witnessing disrespectful and harmful behaviors among peers comparing baseline and follow up mean scores on a scale assessing likelihood of trying to stop disrespectful behaviors among peers
Change in Recognition of Abuse from Baseline to Follow Up | 3 months after intervention (Time 2), 9 months after intervention (Time 3)
  Recognition of disrespectful and harmful behaviors against girls as abusive comparing baseline and follow up mean scores on the recognition of abusive behavior scale
Change in Gender Equitable Attitudes from Baseline to Follow Up | 3 months after intervention (Time 2), 9 months after intervention (Time 3)
  Assessment of gender-equitable attitudes comparing baseline and follow up mean scores on gender attitudes scale
Change in Condom Use Self-Efficacy from Baseline to Follow Up | 3 months after intervention (Time 2), 9 months after intervention (Time 3)
  Assessment of self-efficacy to use condoms comparing baseline and follow up mean scores on a scale assessing confidence to negotiate condom use
Change in Contraception Attitudes from Baseline to Follow Up | 3 months after intervention (Time 2), 9 months after intervention (Time 3)
  Assessment of attitudes related to contraceptive use comparing baseline and follow up mean scores on a scale assessing contraception attitudes

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh, Division of Adolescent and Young Adult Medicine, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Miller E, Jones KA, Culyba AJ, Paglisotti T, Dwarakanath N, Massof M, Feinstein Z, Ports KA, Espelage D, Pulerwitz J, Garg A, Kato-Wallace J, Abebe KZ. Effect of a Community-Based Gender Norms Program on Sexual Violence Perpetration by Adolescent Boys and Young Men: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2020 Dec 1;3(12):e2028499. doi: 10.1001/jamanetworkopen.2020.28499. PMID 33351083
- [Derived] Miller E, Culyba AJ, Paglisotti T, Massof M, Gao Q, Ports KA, Kato-Wallace J, Pulerwitz J, Espelage DL, Abebe KZ, Jones KA. Male Adolescents' Gender Attitudes and Violence: Implications for Youth Violence Prevention. Am J Prev Med. 2020 Mar;58(3):396-406. doi: 10.1016/j.amepre.2019.10.009. Epub 2019 Dec 27. PMID 31889621
- [Derived] Abebe KZ, Jones KA, Culyba AJ, Feliz NB, Anderson H, Torres I, Zelazny S, Bamwine P, Boateng A, Cirba B, Detchon A, Devine D, Feinstein Z, Macak J, Massof M, Miller-Walfish S, Morrow SE, Mulbah P, Mulwa Z, Paglisotti T, Ripper L, Ports KA, Matjasko JL, Garg A, Kato-Wallace J, Pulerwitz J, Miller E. Engendering healthy masculinities to prevent sexual violence: Rationale for and design of the Manhood 2.0 trial. Contemp Clin Trials. 2018 Aug;71:18-32. doi: 10.1016/j.cct.2018.05.017. Epub 2018 May 23. PMID 29802967